CLINICAL TRIAL: NCT02326948
Title: Alcohol Consumption and Gallbladder Cancer: Case-control Study in Jeju Island, Korea.
Brief Title: Alcohol Consumption and Gallbladder Cancer
Status: Completed | Type: Observational
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Byung Hyo Cha, MD, Director of Digestive Disease Center, Cheju Halla General Hospital
Other Study IDs: 2014-L04
Record Dates: First submitted 2014-12-19; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Gallbladder Cancer
Keywords: Gallbladder cancer; Case-control study; Risk factor; Alcohol consumption; Polypoid lesions of gallbladder; Biliary stone
MeSH Terms: conditions — Gallbladder Neoplasms; Alcohol Drinking; Cholecystolithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gallbladder cancer case group: Gallbladder cancer case group was defined as newly diagnosed gallbladder cancer diagnosed as GBC at the Department of Internal Medicine in Cheju Halla General Hospital, Jeju, Korea from 2009 to 2013.
- Age and sex matched control group: Age and sex matched control group was determined as age-sex matched subjects selected from the participants of Health Promotion Center in the same institute from 2009 to 2012.

SUMMARY:
This case-control study matched by age and sex was performed to evaluate the region specific risk factors for gallbladder cancer in Jeju island, Korea.

DETAILED DESCRIPTION:
In order to estimate region-specific risk factors for gallbladder cancer (GBC) in Jeju island, Korea the investigators performed a case-control study. Among 124 GBC patients and 7088 health controls, the investigators randomly selected 78 cases and 78 age-sex matched controls (1:1 matching) and compared their demographic features, combined diseases, and personal histories about known risk factors until now.

ELIGIBILITY:
Inclusion Criteria:

* Case group : newly diagnosed gallbladder cancer patients in Digestive Disease Center, Department of Internal Medicine in Cheju Halla General Hospitalduring 2008-2013
* Control group : 1:1 age-sex matched controls underwent health care screening program in Department of Health Promotion Center in Cheju Halla General Hospital for 2008-2012.

Exclusion Criteria:

* Case group Ambiguous diagnosis primary tumor involving common bile duct follow up loss without pathologic confirmation Incomplete clinical records Couldn't be assessed the results of operation or radiologic imaging.
* Control group Cases unavailable for gallbladder imaging (abdominal ultrasonography ,computed tomography, or magnetic resonance imaging) Cases underwent previous cholecystectomy before enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Case group was defined as the patients newly diagnosed GBC at the Digestive Disease Center and Department of Internal Medicine, Cheju Halla General Hospital, Jeju, Korea, during 2008 - 2013. And control groups were determined the randomly 1:1 matched subjects by the age and sex distributions of GBC cases, among the health care check-up examinees visited to Health Promotion Center in the same institute and same periods. Total 78 cases among 124 GBC patients and matched 78 controls from 7088 health check-up examinees were included this study.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with alcohol consumption | Up to 3 years

OTHER OUTCOMES:
Number of participants with biliary stone diseases | Up to 3 year
Number of participants with polypoid lesions of gallbladder | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Byung Hyo Cha, M.D., Principal Investigator — Director of Digestive Disease Center, Department of Internal Medicine, Cheju Halla General Hospital, Korea
Locations (1):
- Cheju Halla General Hopsital, Jeju City, Jeju Special Governing Province, South Korea